CLINICAL TRIAL: NCT04523103
Title: Clinical Study of Artificial Assisted Oocyte Activation Technique in IVF Fertilization Failure
Brief Title: Artificial Assisted Activation Following in Fertilization Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A0728
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Fertilization
Keywords: fertilization failure, oocyte activation, calcium ionophore

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Standard ICSI procedure. The MII oocytes that failed fertilization in IVF cycles were injected with activating sperm.
- A1 assisted activation (Experimental): The MII oocytes that failed fertilization in ICSI cycles were activated in calcium ionophore A23187 activation solution for two times.
  Interventions: Behavioral: Artificial Assisted Activation
- A2 assisted activation (Experimental): Fertilization failure MII oocytes were collected in ICSI cycles. After CaCl2 was injected, the oocytes were transferred into the calcium ionophore A23187 solution for two times.
  Interventions: Behavioral: Artificial Assisted Activation
- A3 assisted activation (Experimental): Fertilization failure MII oocytes were collected in ICSI cycles. Mechanical activation was done for the MII oocytes, and then the oocytes were transferred into the calcium ionophore A23187 solution for two times.
  Interventions: Behavioral: Artificial Assisted Activation

INTERVENTIONS:
Behavioral: Artificial Assisted Activation — Artificial assisted activation represents an effective technique to rescue the fertilization failure.
  Arms: A1 assisted activation; A2 assisted activation; A3 assisted activation

SUMMARY:
Fertilization failure is a common problem in assisted reproductive Technology (ART). The main reason for fertilization failure of conventional IVF fertilization is sperm penetration failure, and the main reason of ICSI is insufficient oocyte activation. Artificial assisted activation may provide an effective technique to rescue fertilization failure. In this study, standard ICSI procedures were applied to save fertilization failure of unfertilized mature oocytes in IVF cycles. The unfertilized mature oocytes after ICSI were activated by calcium ion, or injected with calcium chloride/activated with mechanical stimulated and then transfer to calcium ion to improve fertilization. In this study, different artificial assisted activation methods were used to save the fertilization failure and assess its effective and subsequent embryo development potential.

DETAILED DESCRIPTION:
A variety of mechanical, electrical, and chemical methods has been used to trigger the calcium oscillations to activate oocytes. Mechanical and chemical activation are the most commonly used methods for artificial oocyte activation, which can mimic calcium oscillations saving fertilization failure.

Control group, a single spermatozoon was injected into the failed fertilization MII oocyte in conventional IVF cycle. What to do when ICSI fails? The investigators collected the unfertilized MII oocytes and divided them into 3 groups to perform different activation methods, including chemical calcium ionophore activation (experiment group 1), CaCl2 injected combined with calcium ionophore activation (experiment group 2), and mechanical stimulation combined with calcium ionophore activation (experiment group 3). Calcium ionophore A23187 (Sigma) was used for assisted activation. The final solution was 10 μmol/L. The oocytes were exposed to the calcium ionophore A23187 for 10 min at 37°C in 5% CO2. The oocytes were checked for pronucleus formation at 16-20 hours after activation. Fertilized oocytes were cultured in vitro for 3-5 days, the developmental potential of the activated embryos were observed.

This study want to explore the effective of different artificial assisted activation methods, to improve the fertilization outcome of unfertilized oocytes after ICSI or IVF.

ELIGIBILITY:
Inclusion Criteria:

* 8 ≤ Number of retrieved oocytes ≤ 20;
* 18.5< Body Mass Index (BMI) <25;
* The patients who suffered complete fertilization failure or low fertilization after performing standard ICSI/IVF cycle. Low fertilization was defined as less than 33% fertilization rate.

Exclusion Criteria:

* Normal fertilization IVF/ICSI cycle.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
the normal fertilization rate | 12 months
  Fertilization (2PN rate)

SECONDARY OUTCOMES:
the good-quality embryo rate | 12 months
  Embryo quality
the blastocyst formation rate | 12 months
  Embryo quality
the good quality blastocyst rate | 12 months
  Embryo quality

CONTACTS AND LOCATIONS:
Overall Officials: Li Bo, Doctor, Study Chair — Reproductive Medicine Center, Tangdu Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China